CLINICAL TRIAL: NCT06801431
Title: A Pilot Study on the Tolerance, Feasibility, and Impact of Transcutaneous Spinal Cord Stimulation on Bowel Management in Individuals with Motor Complete Spinal Cord Injury Receiving Inpatient Care
Brief Title: Transcutaneous Spinal Cord Stimulation for Bowel Management in Individuals with Motor Complete Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Alexander Whelan, Assistant professor, Physical Medicine and Rehabilitation, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56432
Record Dates: First submitted 2025-01-20; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Neurogenic Bowel; Spinal Cord Injuries (SCI)
Keywords: neurogenic bowel; transcutaneous spinal stimulation
MeSH Terms: conditions — Neurogenic Bowel; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: all patients will be treated with the transcutaneous spinal cord stimulation to see if it affects bowel movements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcutaneous spinal cord stimulation (Experimental): Individuals with motor complete cervicothoracic spinal cord injury admitted to tertiary inpatient rehabilitation
  Interventions: Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — Individuals will receive a 10-day course of daily, 30-minute sessions of transcutaneous spinal cord stimulation to the thoracolumbar spine cord using the Chattanooga Mobile 2 Stim Device. These sessions will be conducted in the morning before bowel care and therapy. Cathode pads will be placed between the T10 and T11 spinous processes and the T12 and L1 spinous processes. Anode pads will be placed over the iliac crests. Stimulation will consist of 1 millisecond duration, biphasic pulses, at 30 Hertz frequency. The intensity of the current, will be adjusted to be suprasensory and sub-motor, and no more than 140 milli-amperes.

SUMMARY:
The primary goals of this pilot trial are to understand the feasibility and safety of thoracolumbar transcutaneous spinal cord stimulation for neurogenic bowel management in individuals with new onset, traumatic, cervicothoracic spinal cord injury admitted to inpatient rehabilitation.

The secondary goal is to understand the clinical impact of thoracolumbar spinal cord stimulation on bowel function.

Study participants will receive a 10-day course of transcutaneous spinal cord stimulation at T10-T11 and T12-L1. Each daily treatment will consist of 30 minutes of stimulation.

Feasibility will be evaluated by documenting how many stimulation sessions were attended per participant, and the average duration of stimulation provided per session (with a maximum value of 30 minutes). It is believed that transcutaneous spinal cord stimulation will be feasible to deliver for participants receiving inpatient rehabilitation.

Safety will be evaluated by documenting hemodynamic parameters (heart and blood pressure) and pain levels during each stimulation session. The skin will be evaluated after treatment to ensure no pressure injuries. Participants will be asked to document bladder continence before and after the two-week stimulation protocol, to understand if there are any changes on bladder function, given similar nerve root innervation as bowel function. Investigators expect that transcutaneous spinal cord stimulation will be safe, with minimal adverse effects on heart, blood pressure, skin integrity, pain levels and bladder continence.

The impact on bowel function will be evaluated by completing a bowel diary documenting the time spent on bowel care per day per participant. Participants will also rate their satisfaction with bowel care before, immediately after and two weeks after the 10-day stimulation protocol. Peak cough flow will be collected before, immediately after and two weeks after the 10-day stimulation protocol, as surrogate measures of abdominal strength, which is important for timely bowel evacuation. It is believed that transcutaneous spinal cord stimulation will reduce time spent on bowel care and improve participant-reported satisfaction with bowel care, and it will be associated with improvements in peak cough flow.

ELIGIBILITY:
Inclusion Criteria:

1. Individual must have a T10 and above AIS A-B traumatic spinal cord injury
2. Individual must be 16 years or older
3. They must be willing to comply with the study procedure and be medically stable
4. They must be at least 3 months since their injury, to minimize the chances that they are in spinal shock, which may influence the impact of TSCS as the peripheral nerves may be less excitable)
5. There must not be any changes to their bowel medications or bowel regimen in the week leading up to the intervention, to minimize any confounding effect on bowel habits
6. They must have bowel care either daily or q2 days

Exclusion Criteria:

1. Individuals with a pacemarker, cochlear implant, baclofen pump or other implantable device that may be affected by electrical stimulation.
2. Individuals with epilepsy
3. Individuals with open wounds at stimulation sites
4. Individuals with implanted metal in the trunk and spinal cord at the cathode pad application sites (i.e. T10 to L2)
5. Individuals with a severe acute medical issue that is felt to affect participation at the discretion of the research team, including individuals with uncontrolled autonomic dysreflexia
6. Individuals who are pregnant or planning to become pregnant, and who may be breastfeeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: number of stimulation sessions attended | From start to end of treatment at 2 weeks
  Feasibility will be calculated as the number of sessions (out of 10) when participants were able to engage in transcutaneous spinal cord stimulation. The reason for missed sessions will be recorded.
Feasibility: duration of stimulation tolerated per session | From start to end of treatment at 2 weeks
  Feasibility will be calculated as the average duration of transcutaneous spinal cord stimulation tolerated by participants each session (i.e. the maximum value is 30 minutes, which is a full session of stimulation)
Blood Pressure | From start to end of each stimulation treatment
  Systolic and diastolic blood pressure will be taken immediately before each stimulation session, every 10 minutes during the 30-minute session, and after completion of each session
Heart rate | From start to end of each stimulation treatment
  Heart rate will be taken immediately before each stimulation session, every 10 minutes during the 30-minute session, and after completion of each session
Pain levels | At the end of each stimulation session
  Participants will be asked to rate their average pain during each session of stimulation (numerical rating scale from 0-10, 10 being maximum pain)
Bladder continence | prior to the start of stimulation period and at the end of stimulation period
  Participants will be asked to document bladder continence immediately before and after finishing 10 days of stimulation, using the Revised Urinary Incontinence scale. This scale is a validated 5 question tool to evaluate urinary continence, with the score ranging from 0 to 15, with higher scores indicative of more distressing incontinence.
Skin health | At the start and end of each stimulation session
  The incidence of pressure injuries with visualization using NPIAP staging, with documentation of size (width and length) will be documented. The skin overlying the cathodes and anodes will be visually inspected before and after each stimulation session.

SECONDARY OUTCOMES:
Time spent on bowel care | One week before the stimulation protocol to two weeks after the stimulation protocol
  Nurses assigned to patient care will complete a bowel diary, which is part of clinical care. This will document the time spent on bowel care, starting one week before TSCS and extending to two weeks after TSCS. The time spent will be calculated from the time of suppository insertion/rectal touch until clean-up by nursing.
Satisfaction with Bowel Care | Before, immediately after and two weeks after the stimulation protocol
  We will have participants rate their satisfaction with bowel emptying before, immediately after and two weeks after TSCS. This will be completed using a numerical rating scale from 0-10, where 0 = no satisfaction and 10 = complete satisfaction.
Peak cough flow | Before, immediately after and two weeks after the stimulation protocol
  We will collect the peak cough before, immediately after the stimulation protocol and 2 weeks after the stimulation protocol. The peak cough flow will be the average of three attempts at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Whelan, MD, Principal Investigator — NSHA

IPD SHARING:
Plan to Share IPD: No